CLINICAL TRIAL: NCT00147017
Title: Regulation of the Release of Inflammatory Mediators From Lung Macrophages.
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Novartis (Industry); Boehringer Ingelheim (Industry); Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 01-093; DHTAB PN1257; DHTAB PC3608; DHTAB P00134
Record Dates: First submitted 2005-09-05; First posted 2005-09-07 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-11

CONDITIONS: COPD; Chronic Bronchitis; Emphysema
Keywords: macrophage; inflammation; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema; Inflammation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — protein samples have been retained
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Smokers: All subjects had a smoking history of >15 pack years
- Ex-smokers: Ex-smokers had ceased smoking for >6 months.
- Emphysema lung transplant: The emphysema subjects were all undergoing lung transplants.

SUMMARY:
The aim of this study is to investigate the mechanisms whereby specific white cells called macrophages found in the lung release inflammatory mediators or chemicals together with enzymes that destroy the surrounding lung tissue. The hypothesis is that in diseases such as chronic obstructive pulmonary disease (COPD), lung macrophages release either more or different types of inflammatory mediators and/or destructive enzymes compared to subjects without COPD. We will isolate macrophages from small pieces of lung parenchyma. These samples are derived from lobes resected for carcinoma of the lung. We would aim to examine the responses of tissue derived macrophages in three groups of subjects, namely (i) non-smoking controls (lung carcinoma as secondary metastasis), (ii) smokers without clinical or histological signs of COPD and (iii) smokers with COPD. The resected lung tissue will be cut into small pieces and washed in order to release the macrophages from the tissue. The macrophages will then be isolated from other cell types in the washings. We will then use these isolated cells in vitro to examine the cell surface receptors in order to compare these macrophage cells with macrophages reported from bronchoalveolar lavage and monocyte derived macrophage models. We will then examine inflammatory mediator synthesis and release following stimulation of these cells. We will also examine the regulation and release of enzymes known to damage lung tissue. Using these two models we will then examine the signal transduction pathways that lead to this activation of the macrophages and investigate the effects of novel therapeutic agents to inhibit inflammatory mediator and/or enzyme synthesis and release. The objective is to identify the mechanisms whereby macrophages respond to pro-inflammatory conditions seen in COPD with a view to identify novel targets for drug therapy.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is the fifth leading cause of death in the UK and is the only common cause of death that is increasing. COPD is currently 6th in the global impact of diseases and is predicted to by the 3rd leading cause of death by 2020. In the UK for 2000-2001 the estimated cost of COPD related illness is estimated at ~£980 million of which pharmacotherapy accounts for 48% of expenditure. At present pharmacotherapy for COPD is purely symptomatic with no drugs currently available that can halt the relentless progression of this disease. Therefore, there is a need for improved therapy for the treatment of COPD. Cigarette smoking is the major risk factor in the development of COPD, yet for reasons unknown only ~15% of smokers develop this disease, suggesting there is an underlying genetic component.

COPD encompasses chronic bronchitis, small airways disease and emphysema and is associated with increased inflammatory cells in the lung including neutrophils, macrophages and CD8+ T-lymphocytes. This inflammatory infiltrate is thought to be responsible for all the pathophysiological features of COPD but the precise mechanisms underlying this inflammatory response are unknown.In particular the macrophage is thought to mediate all the pathophysiological features of this disease. To this end, macrophages will be isolated from lung parenchyma using discontinuous percoll gradients. The cells will then be cultured overnight prior to assessment of inflammatory mediator release. Cells will be stimulated by a variety of agents including but not exclusively LPS, IL-1beta or TNF-alpha. The release of inflammatory mediators into the cell culture media will be measured using ELISA techniques. Enzyme activity will also be measured in both the cells and the culture media. Cell surface expression of specific markers will be assessed using immunocytochemistry and FACS analysis. Function of macrophages will be assessed by measuring phagocytotic activity by FACS analysis and fluorimetry. Specific signal transduction pathways will be assessed by the use of specific pathway inhibitors and gene expression measured by real-time PCR. The effects of novel therapeutic agents will be tested on these outputs with the aim to identify novel therapies for COPD.

ELIGIBILITY:
Inclusion Criteria:

- All subjects undergoing surgical resection of the lung

Exclusion Criteria:

- Anyone unable to understand the consent form

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects undergoing lung resection surgery
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2001-06 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louise E Donnelly, PhD, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton Hospital/NHLI Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Smith SJ, Fenwick PS, Nicholson AG, Kirschenbaum F, Finney-Hayward TK, Higgins LS, Giembycz MA, Barnes PJ, Donnelly LE. Inhibitory effect of p38 mitogen-activated protein kinase inhibitors on cytokine release from human macrophages. Br J Pharmacol. 2006 Oct;149(4):393-404. doi: 10.1038/sj.bjp.0706885. Epub 2006 Sep 4. PMID 16953188

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Smokers | Ex-smokers | Emphysema Lung Transplant
Started | 6 | 7 | 4
Completed | 6 | 7 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Smokers | Ex-smokers | Emphysema Lung Transplant | Total
Number analyzed (Participants) | 6 | 7 | 4 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (3.2) | 52.3 (3.7) | 52.0 (0.8) | 53.4 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 1 | 8
  Male | 3 | 3 | 3 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 7 | 4 | 17
Smoking history [Mean (Standard Deviation); unit: pack/years] | 34.3 (8.4) | 41.0 (16.3) | NA (NA) — Data is not available from the transplant team | 37.9 (12.3)
FEV1 (% predicted) [Mean (Standard Deviation); unit: % predicted] | 87.9 (6.1) | 83.2 (3.5) | NA (NA) — Data was not available from the transplant team | 85.4 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Macrophage Activation, TNF-a
Description: measure release of inflammatory mediators from isolated macrophages
Time Frame: 20 hours
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Smokers | Ex-smokers | Emphysema Lung Transplant
Number analyzed (Participants) | 6 | 7 | 4
ng/ml | 6.1 (2.2) | 3.8 (1.5) | 2.6 (1.2)
Statistical Analysis 1: Comparison: Smokers vs Ex-smokers vs Emphysema Lung Transplant; Test type: Superiority; p = 0.05, Kruskal-Wallis — calculated

2. Primary Outcome: Macrophage Activation, GM-CSF
Description: GM-CSF, granulocyte macrophage-colony stimulating factor
Time Frame: 20 hours
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Smokers | Ex-smokers | Emphysema Lung Transplant
Number analyzed (Participants) | 6 | 7 | 4
ng/ml | 2.2 (0.5) | 1.8 (0.5) | 2.6 (1.2)
Statistical Analysis 1: Comparison: Smokers vs Ex-smokers vs Emphysema Lung Transplant; Test type: Superiority; p = 0.05, Kruskal-Wallis — calculated

3. Primary Outcome: Interleukin, IL-8
Time Frame: 20 hours
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Smokers | Ex-smokers | Emphysema Lung Transplant
Number analyzed (Participants) | 6 | 7 | 4
ng/ml | 220.8 (67.1) | 251.2 (58.7) | 167.8 (49.5)
Statistical Analysis 1: Comparison: Smokers vs Ex-smokers vs Emphysema Lung Transplant; Test type: Superiority; p = 0.05, Kruskal-Wallis — calculated

ADVERSE EVENTS:
Time Frame: 20 hours
Arm/Group | Smokers | Ex-smokers | Emphysema Lung Transplant
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 0/4
Other Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes